CLINICAL TRIAL: NCT02907242
Title: Revealed Versus Concealed Criteria for Placental Insufficiency in Unselected Obstetric Population in Late Pregnancy: a Multicenter Randomized Controlled Trial
Brief Title: Revealed Versus Concealed Cerebroplacental Ratio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francesc Figueras, Obstetrics Department Head Hospital Clinic Barcelona, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RATIO37
Record Dates: First submitted 2016-08-01; First posted 2016-09-20 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Stillbirth
Keywords: stillbirth; cerebroplacental ratio; fetal growth restriction
MeSH Terms: conditions — Stillbirth; Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concealment (No Intervention): Cerebroplacental ratio measurement at 37 weeks of pregnancy only taken into account if estimated fetal weight <p10
- Revealment (Other): Cerebroplacental ratio measurement at 37weeks and labor induction in case of cerebroplacental ratio <p5
  Interventions: Other: Revealment

INTERVENTIONS:
Other: Revealment — Cerebroplacental ratio revealment
  Arms: Revealment

SUMMARY:
The purpose of this study is to evaluate the role of an integrated strategy at selecting fetuses for delivery at term based on a combination of fetal biometry and cerebroplacental ratio (CPR) to reduce stillbirth rate and adverse perinatal outcome.

DETAILED DESCRIPTION:
This is a multicenter, open-label randomized trial with groups in parallel. Singleton pregnancies are recruited after routine second trimester scan (19+0 to 22+6 weeks of gestation) and randomly allocated at that moment to revealed or concealed strategy. A routine scan will be booked at 36-37 weeks. For a reduction of the stillbirth rate of 3‰ (from 5‰ to 2‰), assuming a type I error of 5% and aiming for a power of 80% a total of 11,582 subjects (5791 per arm) were projected. The participating centers sum up 12,000 deliveries a year. It is not possible to blind participants, obstetricians, or outcome assessors to the study group.

General hypothesis: A proportion of fetuses with "normal" growth as per current standards have placental insufficiency and restriction of their growth potential. These fetuses exhibit biophysical changes expressed by abnormal cerebroplacental ratio. A combination of this marker with fetal biometry for the detection of fetuses affected by fetal growth restriction could identify a group of babies on which labor induction once term is reached may prevent the occurrence of adverse outcomes.

Specific hypothesis

* The cerebroplacental ratio has predictive value in late pregnancy for placental insufficiency.
* The cerebroplacental ratio could improve the effectiveness of late pregnancy screening for the prediction placental insufficiency-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Viable singleton non-malformed fetus
* Available first-trimester US dating
* Maternal age at recruitment ≥18 years
* No adverse medical or obstetrical history at booking
* Capacity to give informed consent

Exclusion Criteria:

* Abnormal karyotype
* Structural abnormalities
* Congenital infections

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11582 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Stillbirth | between 37 and 42 weeks of pregnancy
  Perinatal death

SECONDARY OUTCOMES:
Adverse perinatal outcome | Up to 28 days after delivery
  Severe neurological and non-neurological adverse outcome
Fetal Growth Restriction Detection | 3 years
  To detect prenatal low birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Gratacos, PhD, Study Chair — Hospital Clinic
Locations (9):
- Hospital Clínico Universitario de Santiago de Chile, Santiago, Chile
- Czechia (2):
  - Palacky University Hospital, Olomouc
  - Ladislav Krofta, Prague
- Eyal Zohav, Tel Aviv, Israel
- Hospital de Querétaro, Querétaro, Mexico
- Anna Kajdy, Warsaw, Poland
- Spain (3):
  - Hospital Clinic, Barcelona
  - Elena Escazzocchio, Barcelona
  - Elena Ferriols Perez, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rial-Crestelo M, Lubusky M, Parra-Cordero M, Krofta L, Kajdy A, Zohav E, Ferriols-Perez E, Cruz-Martinez R, Kacerovsky M, Scazzocchio E, Roubalova L, Socias P, Haslik L, Modzelewski J, Ashwal E, Castella-Cesari J, Cruz-Lemini M, Gratacos E, Figueras F; RATIO37 Study Group. Term planned delivery based on fetal growth assessment with or without the cerebroplacental ratio in low-risk pregnancies (RATIO37): an international, multicentre, open-label, randomised controlled trial. Lancet. 2024 Feb 10;403(10426):545-553. doi: 10.1016/S0140-6736(23)02228-6. Epub 2024 Jan 11. PMID 38219773
- [Derived] Figueras F, Gratacos E, Rial M, Gull I, Krofta L, Lubusky M, Cruz-Martinez R, Cruz-Lemini M, Martinez-Rodriguez M, Socias P, Aleuanlli C, Cordero MCP. Revealed versus concealed criteria for placental insufficiency in an unselected obstetric population in late pregnancy (RATIO37): randomised controlled trial study protocol. BMJ Open. 2017 Jun 15;7(6):e014835. doi: 10.1136/bmjopen-2016-014835. PMID 28619771